CLINICAL TRIAL: NCT02357173
Title: A Trial of E-cigarettes: Natural Uptake, Patterns and Impact of Use
Brief Title: A Trial of E-cigarettes in Current Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00035634; 1R21DA037407-01 (NIH)
Record Dates: First submitted 2014-10-03; First posted 2015-02-06 (Estimated); Results first posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2016-11

CONDITIONS: Smoking; Nicotine Dependence; Nicotine Dependence, Other Tobacco Product
Keywords: smoking; nicotine; tobacco products; electronic cigarette
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cigarette group (Active Comparator): This group (1/3 of the sample) will not receive electronic cigarettes to sample and will continue smoking their regular cigarettes as much or as little as they would like.
  Interventions: Other: cigarette group
- electronic cigarette (Experimental): This group (2/3 of the sample) will be given electronic cigarettes for a 3-week period, to use as much or as little as they would like.
  Interventions: Other: electronic cigarette

INTERVENTIONS:
Other: electronic cigarette
  Other Names: Blu ecigs
  Arms: electronic cigarette
Other: cigarette group
  Arms: cigarette group

SUMMARY:
The purpose of this study is to examine cigarette smokers' use of electronic cigarettes (e-cigarettes), and how use of e-cigarettes affects short term smoking behavior.

DETAILED DESCRIPTION:
Study initiation will commence after the first telephone contact (phone pre-screen), at the baseline visit. Additional lab visits will occur at days 8, 15, and 22 (visits 2-4). At the first study visit, 2/3rds of the participants will be randomly assigned to sample e-cigarettes and 1/3rd will not. Participants in the e-cigarette group will be provided with sufficient product to sample and use as they wish, but with minimal instruction on purpose and level of use (non-use is an outcome). Smokers in the control group will smoke their own brand of cigarettes, as they wish, for the duration of the sampling period. All participants will engage in ecological momentary assessments, which will be completed 3 times daily for 3 weeks. In-person follow-up assessments will be conducted at 1, 2, and 3 months after the final lab visit (Day 22).

Overall, each participant will be contacted 8 times: at the phone pre-screening, the 4 lab visits, and 3 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* current smoker of at least 5 cigarettes per day for at least 1 year
* at least some concern for health effects of smoking
* having an easily accessible email address

Exclusion Criteria:

* past six month use of any e-cigarette
* lifetime ever purchase of any e-cigarette
* recent history of cardiovascular distress (heart attack in past year; arrhythmia; uncontrolled hypertension)
* recent history (past 3 months) of Chronic Obstructive Pulmonary Disease (COPD), cancer (any non-dermatologic), or uncontrolled diabetes mellitus
* pregnant or breastfeeding
* any major current psychiatric impairment, including current alcohol/drug abuse/dependence
* use of non-cigarette tobacco products (e.g., cigarillos) in the last 30 days
* current use of any smoking cessation medications
* current enrollment in a smoking cessation treatment study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Carpenter, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 16 mg Electronic Nicotine Delivery Systems (ENDS); 24 mg Electronic Nicotine Delivery Systems (ENDS): Study Participants were randomized in a 2:1 ratio to receive electronic nicotine delivery systems (ENDS) or not.
  Changes in product design, i.e., improved nicotine delivery (16mg vs. 24mg), midway through the study allowed the unexpected but compelling opportunity to examine two ENDS products compared to control group.
- Control Group: This group (1/3 of the sample) did not receive electronic cigarettes to sample and continued smoking their regular cigarettes as much or as little as they chose.
Period: Overall Study
Arm/Group | 16 mg Electronic Nicotine Delivery Systems (ENDS) | 24 mg Electronic Nicotine Delivery Systems (ENDS) | Control Group
Started | 25 | 21 | 22
Completed | 19 | 15 | 16
Not Completed | 6 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 16 mg Electronic Nicotine Delivery Systems (ENDS) | 24 mg Electronic Nicotine Delivery Systems (ENDS) | Control Group | Total
Number analyzed (Participants) | 25 | 21 | 22 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (14.4) | 40.9 (12.3) | 42.3 (14.2) | 42.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 14 | 41
  Male | 7 | 12 | 8 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 14 | 10 | 13 | 37
  Race: Black or African American | 10 | 11 | 9 | 30
  Race: Multiracial | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 21 | 22 | 68

OUTCOME MEASURES:

1. Primary Outcome: Uptake of Electronic Nicotine Delivery Systems (ENDS)
Description: % of participants by group used e-cigarettes in week 16
Time Frame: study week 16
Measure: Number; unit: percentage of participants
Arm/Group | 24 mg Electronic Nicotine Delivery Systems (ENDS) | 16 mg Electronic Nicotine Delivery Systems (ENDS) | Control Group
Number analyzed (Participants) | 21 | 25 | 22
percentage of participants | 57.14 | 32 | 13.64

2. Primary Outcome: Independent Purchase of an ENDs Product
Description: % of participants by group who purchased an ENDs product on their own during the study
Time Frame: study enrollment to study week 16
Measure: Number; unit: percentage of participants
Arm/Group | 24 mg Electronic Nicotine Delivery Systems (ENDS) | 16 mg Electronic Nicotine Delivery Systems (ENDS) | Control Group
Number analyzed (Participants) | 21 | 25 | 22
percentage of participants | 57 | 28 | 14

3. Primary Outcome: % Quit Attempts
Description: % of participants who made any quit attempt during study
Time Frame: study enrollment to study week 16
Measure: Number; unit: percentage of participants
Arm/Group | 24 mg Electronic Nicotine Delivery Systems (ENDS) | 16 mg Electronic Nicotine Delivery Systems (ENDS) | Control Group
Number analyzed (Participants) | 21 | 25 | 22
percentage of participants | 47.6 | 40 | 27.3

4. Primary Outcome: Point Prevalence Abstinence
Description: % of participants with CO-verified cigarette abstinence at study week 16
Time Frame: week 16
Measure: Number; unit: percentage of participants
Arm/Group | 24 mg Electronic Nicotine Delivery Systems (ENDS) | 16 mg Electronic Nicotine Delivery Systems (ENDS) | Control Group
Number analyzed (Participants) | 21 | 25 | 22
percentage of participants | 9.5 | 4.0 | 4.6

ADVERSE EVENTS:
Time Frame: study week 2 to study week 16
Arm/Group | 24 mg Electronic Nicotine Delivery Systems (ENDS) | 16 mg Electronic Nicotine Delivery Systems (ENDS) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 11/21 | 9/25 | 8/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24 mg Electronic Nicotine Delivery Systems (ENDS) (N=21) | 16 mg Electronic Nicotine Delivery Systems (ENDS) (N=25) | Control Group (N=22)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (7) | 4 (6)
nausea (Gastrointestinal disorders) | 5 (6) | 3 (3) | 4 (4)
headache (Nervous system disorders) | 3 (3) | 1 (1) | 4 (7)
Mouth/throat irritation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (5)
Trouble sleeping (General disorders) | 1 (1) | 1 (1) | 3 (4)
heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
dizziness or lightheadness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
other (General disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
* small sample size
* 1st generation e-cigarette device
* no placebo group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No